CLINICAL TRIAL: NCT06370091
Title: Effect of Xylitol-based Chewing Gums, Sugar-free and Sugared, on Salivary Flow and pH in Young Adults: Randomized Controlled Clinical Trial
Brief Title: Effect of Xylitol-based Chewing Gums, Sugar-free and Sugared, on Salivary Flow and pH in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica de Cuenca (Other)
Responsible Party: Principal Investigator, Miriam Lima, Doctor in Stomatological Sciences, Universidad Católica de Cuenca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PICVII19-41
Record Dates: First submitted 2024-04-06; First posted 2024-04-17 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-11

CONDITIONS: Healthy
Keywords: Chewing gum; Xylitol; Sugars; Salival; Dental Plaque
MeSH Terms: conditions — Dental Plaque | interventions — Paraffin

STUDY DESIGN:
Intervention Model Description: It will be an experimental study through a double-blind parallel randomized controlled trial.
  All saliva samples will be collected using the spitting method. Each participant will provide a basal saliva sample for 5 minutes. Participants must meet the following inclusion criteria: having at least 20 teeth, providing written informed consent, and being willing to comply with the study procedures. The exclusion criteria will include individuals with systemic, infectious, or inflammatory diseases or those taking medications, antibiotics, or fluoride in the last month; regular consumers of products and mouthwashes containing xylitol or sorbitol, with abnormal salivary flow (<1 ml/min), pregnant women or those on contraceptive pill treatment, or with abnormal dietary habits; subjects with periodontal disease or presence of dental caries
Who Masked: Participant, Investigator
Masking Description: Participants who meet the selection criteria will be probabilistically assigned using simple random sampling through a lottery system. An urn will be used to draw colors corresponding to a type of chewing gum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- G1: Gum of Xylitol (Experimental): They will consume chewing gum with xylitol (Xylichew), and stimulated saliva will be collected at three time intervals: T2 from 5 to 10 minutes, T3 from 15 to 20 minutes, and T4 from 25 to 30 minutes after the start of chewing gum consumption
  Interventions: Other: Gum of Xylitol
- G2: Gum of sugar free (Active Comparator): They will consume sugar-free chewing gum (Trident), and stimulated saliva will be collected at three time intervals: T2 from 5 to 10 minutes, T3 from 15 to 20 minutes, and T4 from 25 to 30 minutes after the start of chewing gum consumption
  Interventions: Other: Gum of sugar free
- G3: Gum of sugar (Active Comparator): Formed by participants who will chew sugared gum (Agogó), and stimulated saliva will be collected at three time intervals: T2 from 5 to 10 minutes, T3 from 15 to 20 minutes, and T4 from 25 to 30 minutes after the start of chewing gum consumption
  Interventions: Other: Gum of sugar
- G4: paraffin wax (Placebo Comparator): The control group will chew paraffin wax (Dentek), and stimulated saliva will be collected at three time intervals: T2 from 5 to 10 minutes, T3 from 15 to 20 minutes, and T4 from 25 to 30 minutes after the start of chewing paraffin wax
  Interventions: Other: Paraffin wax

INTERVENTIONS:
Other: Gum of Xylitol — After each sample, the salivary pH level will be measured, and the amount of basal saliva will be weighed. This amount will be subtracted from the accumulated saliva at T4 to establish salivary flow
  Arms: G1: Gum of Xylitol
Other: Gum of sugar free — After each sample, the salivary pH level will be measured, and the amount of basal saliva will be weighed. This amount will be subtracted from the accumulated saliva at T4 to establish salivary flow
  Arms: G2: Gum of sugar free
Other: Gum of sugar — After each sample, the salivary pH level will be measured, and the amount of basal saliva will be weighed. This amount will be subtracted from the accumulated saliva at T4 to establish salivary flow
  Arms: G3: Gum of sugar
Other: Paraffin wax — After each sample, the salivary pH level will be measured, and the amount of basal saliva will be weighed. This amount will be subtracted from the accumulated saliva at T4 to establish salivary flow
  Arms: G4: paraffin wax

SUMMARY:
This study was planned to evaluate the effects of xylitol-based chewing gums, sugar-free and sugared, on salivary flow and pH in young adults.

DETAILED DESCRIPTION:
Chewing gum stimulates salivary flow, neutralizes and raises pH, and serves as a medium for administering therapeutic agents. However, global increases in sugar consumption have led to the development of chewing gums containing sugar substitutes, including polyols or non-fermentable sugars, of which the most commonly used are nutritive sweeteners such as sorbitol and xylitol.The use of polyol-containing chewing gums could play a role in preventing dental caries compared to not using gum or using sugared gum, most likely due to increased salivary flow and pH, improving enamel lesion remineralization; however, xylitol has anticariogenic properties influencing the reduction of dental plaque.

The study will conduct as a prospective randomized controlled trial. The population will consist of all enrolled students (1275 students) in the Dentistry program at the Catholic University aged 18 to 25 who voluntarily meet the inclusion criteria. The sample size will be 21 participants in each group, but it will be adjusted for a 15% loss of information or study dropout, thus requiring 25 participants in each group. Participants who meet the selection criteria will be probabilistically assigned using simple random sampling through a lottery system to four groups: the first group (G1) will consume xylitol chewing gum, the second group (G2) will consume sugar-free gum, the third group (G3) will consume sugared gum, and the fourth group (G4), the control, will chew paraffin.

Saliva samples will be taken between 8 to 10 am, taking into account that subjects should not have ingested food, smoked, or brushed their teeth at least 1 hour prior to sample collection. They will be asked to rinse their mouth with pure water to remove any food residue. Subsequently, they will be seated in a chair in an upright position with the head slightly tilted forward and eyes open, and the basal saliva sample will be taken as indicated by the established protocol of the collection method for unstimulated saliva by Tomas Seif. Before starting the test, they will be asked to swallow saliva, keep their mouth slightly open, and allow saliva to drain into the tube. The test lasts for five minutes and the salivary pH will be evaluated and recorded, labeled as T1. For stimulated saliva, the protocol dictated by the Faculty of Dentistry at the University of Southern California will be used. Through the drainage method, stimulated saliva will be collected in another pre-weighed test tube at three more time intervals: T2 from 5 to 10 minutes, T3 from 15 to 20 minutes, and T4 from 25 to 30 minutes after starting chewing gum consumption. The Measurement of saliva pH level will be evaluated immediately using a pH meter (BT-675 meter, Boeco-Germany), while the salivary flow will be evaluated by the difference in weight of the basal pH with the final pH.

Data will be entered into an Excel spreadsheet and data analysis will be performed. The analysis will be conducted using SPSS v.25, with descriptive data analysis. Chi-square test will be used for demographic data, Levene's test will determine data homogeneity, and ANOVA will determine differences in means, followed by Tukey's post-hoc comparison to find significant differences between group means, with a significance level of p<0.05.

The expected results, that the mean salivary pH and flow will differ among the different chewing gums

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet at least 20 teeth.
* Providing written informed consent. and being willing to comply with the study procedures.
* Being willing to comply with the study procedures

Exclusion Criteria:

* Individuals with systemic, infectious, or inflammatory diseases
* Individuals who are taking medications, antibiotics, or fluoride in the last month.
* Regular consumers of products and mouthwashes containing xylitol or sorbitol.
* Individuals with abnormal salivary flow (<1 ml/min).
* Pregnant women or those on contraceptive pill treatment.
* Individuals with abnormal dietary habits.
* Subjects with periodontal disease or presence of dental caries.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
G1: Gum of xilytol | The trial period for each participant is 35 minutes in total. Salivary pH at 10 minutes, salivary pH at 20 minutes, salivary pH at 30 minutes. Basal salivary volume and salivary volume at 35 minutes.
  Measurement of basal salivary pH (T1), salivary pH at T2, salivary pH at T3, salivary pH at T4. Each Falcon tube will be weighed empty, with basal saliva, and at time T4, and then the difference will be established to determine salivary flow.
G2: Gum of sugar free | The trial period for each participant is 35 minutes in total. Salivary pH at 10 minutes, salivary pH at 20 minutes, salivary pH at 30 minutes. Basal salivary volume and salivary volume at 35 minutes.
  Measurement of basal salivary pH (T1), salivary pH at T2, salivary pH at T3, salivary pH at T4. Each Falcon tube will be weighed empty, with basal saliva, and at time T4, and then the difference will be established to determine salivary flow.
G3: Gum of sugar | The trial period for each participant is 35 minutes in total. Salivary pH at 10 minutes, salivary pH at 20 minutes, salivary pH at 30 minutes. Basal salivary volume and salivary volume at 35 minutes.
  Measurement of basal salivary pH (T1), salivary pH at T2, salivary pH at T3, salivary pH at T4. Each Falcon tube will be weighed empty, with basal saliva, and at time T4, and then the difference will be established to determine salivary flow.
G4: Parafinn wax | The trial period for each participant is 35 minutes in total. Salivary pH at 10 minutes, salivary pH at 20 minutes, salivary pH at 30 minutes. Basal salivary volume and salivary volume at 35 minutes.
  Measurement of basal salivary pH (T1), salivary pH at T2, salivary pH at T3, salivary pH at T4. Each Falcon tube will be weighed empty, with basal saliva, and at time T4, and then the difference will be established to determine salivary flow.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Lima, PhD, Principal Investigator — Universidad Católica de Cuenca
Locations (1):
- Miriam Lima, Cuenca, Azuay, Ecuador

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) underlying the results of the publication will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available from July 2024 to January 2025.
Access Criteria: The data will be shared with anyone requesting it via email, stating the purpose of the request

REFERENCES:
- [Result] Giacaman RA. Sugars and beyond. The role of sugars and the other nutrients and their potential impact on caries. Oral Dis. 2018 Oct;24(7):1185-1197. doi: 10.1111/odi.12778. Epub 2017 Oct 6. PMID 28898520
- [Result] Vantipalli UK, Avula SSJ, Enuganti S, Bandi S, Kakarla P, Kuravadi RV. Effect of three commercially available chewing gums on salivary flow rate and pH in caries-active and caries-free children: An in vivo study. J Indian Soc Pedod Prev Dent. 2017 Jul-Sep;35(3):254-259. doi: 10.4103/JISPPD.JISPPD_256_16. PMID 28762353
- [Result] Shinde MR, Winnier J. Comparative evaluation of Stevia and Xylitol chewing gum on salivary Streptococcus mutans count - A pilot study. J Clin Exp Dent. 2020 Jun 1;12(6):e568-e573. doi: 10.4317/jced.55720. eCollection 2020 Jun. PMID 32665816
- [Result] Rafeek R, Carrington CVF, Gomez A, Harkins D, Torralba M, Kuelbs C, Addae J, Moustafa A, Nelson KE. Xylitol and sorbitol effects on the microbiome of saliva and plaque. J Oral Microbiol. 2018 Oct 23;11(1):1536181. doi: 10.1080/20002297.2018.1536181. eCollection 2019. PMID 30598728
- [Result] Zimmer S, Spyra A, Kreimendahl F, Blaich C, Rychlik R. Elevating the use of sugar-free chewing gum in Germany: cost saving and caries prevention. Acta Odontol Scand. 2018 Aug;76(6):407-414. doi: 10.1080/00016357.2018.1487994. Epub 2018 Jun 27. PMID 29947271
- [Result] Hashiba T, Takeuchi K, Shimazaki Y, Takeshita T, Yamashita Y. Chewing xylitol gum improves self-rated and objective indicators of oral health status under conditions interrupting regular oral hygiene. Tohoku J Exp Med. 2015 Jan;235(1):39-46. doi: 10.1620/tjem.235.39. PMID 25744362
- [Result] Keukenmeester RS, Slot DE, Putt MS, Van der Weijden GA. The effect of medicated, sugar-free chewing gum on plaque and clinical parameters of gingival inflammation: a systematic review. Int J Dent Hyg. 2014 Feb;12(1):2-16. doi: 10.1111/idh.12026. Epub 2013 Jun 24. PMID 23790138
- [Result] Tapiainen T, Renko M, Kontiokari T, Uhari M. Xylitol concentrations in the saliva of children after chewing xylitol gum or consuming a xylitol mixture. Eur J Clin Microbiol Infect Dis. 2002 Jan;21(1):53-5. doi: 10.1007/s10096-001-0654-4. PMID 11913502
- [Result] Navazesh M, Kumar SK; University of Southern California School of Dentistry. Measuring salivary flow: challenges and opportunities. J Am Dent Assoc. 2008 May;139 Suppl:35S-40S. doi: 10.14219/jada.archive.2008.0353. PMID 18460678

DOCUMENTS (1):
  • Study Protocol (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT06370091/Prot_000.pdf